CLINICAL TRIAL: NCT05557955
Title: Predicting Clinical Outcomes Based on Dynamic Breathomics Testing in Esophageal Squamous Cell Carcinoma Receiving Chemoradiotherapy: A Prospective Observational Study (EC-CRT-005)
Brief Title: Identification of Breath Biomarkers in Esophageal Cancer
Acronym: EC-CRT-005
Status: Completed | Type: Observational
Sponsor: Mian XI (Other)
Responsible Party: Sponsor-Investigator, Mian XI, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: B2022-474-01
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Chemoradiotherapy; Dynamic breathomics testing
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant chemoradiotherapy group: All patients will receive standard fractionation radiation therapy (RT) scheme: 40-50.4 Gy in 20-28 fractions over 4-6 weeks using intensity-modulated radiotherapy, concurrently with platinum- or taxane-based chemotherapy, with or without PD-1 inhibitors. All patients will undergo esophagectomy 6-8 weeks after the completion of neoadjuvant CRT. Dynamic breathing testing was performed before, during, and after radiotherapy.
  Interventions: Other: Breathing test
- Definitive chemoradiotherapy group: All patients will receive standard fractionation radiation therapy (RT) scheme: 50-50.4 Gy in 25-28 fractions over 5-6 weeks using intensity-modulated radiotherapy, concurrently with platinum- or taxane-based chemotherapy, with or without PD-1 inhibitors. Dynamic breathing testing was performed before, during, and after radiotherapy.
  Interventions: Other: Breathing test

INTERVENTIONS:
Other: Breathing test — Dynamic breathing testing will be performed before, during, and after radiotherapy. Volatile organic compounds (VOCs) will be collected.

SUMMARY:
Neoadjuvant chemoradiotherapy (CRT) followed by surgery or definitive CRT is the standard treatment for locally advanced esophageal squamous cell carcinoma (ESCC), but the clinical outcomes are not satisfactory. Breathomics testing is a promising, non-invasive, simple method for detection and screening for ESCC. This observational study aimed to role of exhaled volatile organic compounds (VOCs) in predicting the efficacy and risk of recurrence in patients with locally advanced ESCC who received CRT.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (CRT) followed by surgery or definitive CRT is the standard treatment for locally advanced esophageal squamous cell carcinoma (ESCC), but the clinical outcomes are not satisfactory. Breathomics testing is a promising, non-invasive, simple method for detection and screening for ESCC. This observational study aimed to role of exhaled volatile organic compounds (VOCs) in predicting the efficacy and risk of recurrence in patients with locally advanced ESCC who received CRT. All patients will receive standard fractionation radiation therapy (RT) scheme: 40-50.4 Gy in 20-28 fractions over 4-6 weeks using intensity-modulated radiotherapy, concurrently with platinum- or taxane-based chemotherapy, with or without PD-1 inhibitors. All patients will undergo esophagectomy 6-8 weeks after the completion of neoadjuvant CRT. Dynamic breathing testing was performed before, during, and after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Absence of hematogenous metastasis disease, confirmed by endoscopic ultrasound (EUS) and PET-CT scan (according to UICC TNM version 8);
3. Age at diagnosis >18 years;
4. No prior cancer therapy;
5. Estimated life expectancy >6 months;
6. Eastern Cooperative Oncology Group performance status ≤ 2
7. No history of concomitant or previous malignancy;
8. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 4.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 100×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
9. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Patients with hematogenous metastasis disease at diagnosis;
3. Female patients who are pregnant or lactating;
4. Inability to provide informed consent due to psychological, familial, social and other factors;
5. Patients who cannot tolerate chemoradiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia.
6. The physical condition is not enough to provide 0.5L exhalation at one time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 230 patients with ESCC who undergo neoadjuvant chemoradiotherapy or definitive radiotherapy will be included.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
overall survival. | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 24 months.
  A predictive model based on exhaled volatile organic compounds to predict overall survival.

SECONDARY OUTCOMES:
clinical complete response. | 3 months after the treatment (plus or minus 7 days)
  A predictive model based on exhaled volatile organic compounds to predict clinical complete response. Tumor response was evaluated 3 months after the completion of treatment based on CT or PET-CT scans, endoscopy with biopsies. RECIST (Response Evaluation Criteria in Solid Tumors) criteria was used to determine the tumor response.
recurrence. | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  A predictive model based on exhaled volatile organic compounds to predict recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Study Director — Sun Yat-sen University
Locations (1):
- Mian Xi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang P, Huang Q, Meng S, Mu T, Liu Z, He M, Li Q, Zhao S, Wang S, Qiu M. Identification of lung cancer breath biomarkers based on perioperative breathomics testing: A prospective observational study. EClinicalMedicine. 2022 Apr 16;47:101384. doi: 10.1016/j.eclinm.2022.101384. eCollection 2022 May. PMID 35480076
- [Result] Meng S, Li Q, Zhou Z, Li H, Liu X, Pan S, Li M, Wang L, Guo Y, Qiu M, Wang J. Assessment of an Exhaled Breath Test Using High-Pressure Photon Ionization Time-of-Flight Mass Spectrometry to Detect Lung Cancer. JAMA Netw Open. 2021 Mar 1;4(3):e213486. doi: 10.1001/jamanetworkopen.2021.3486. PMID 33783517
- [Result] Markar SR, Wiggins T, Antonowicz S, Chin ST, Romano A, Nikolic K, Evans B, Cunningham D, Mughal M, Lagergren J, Hanna GB. Assessment of a Noninvasive Exhaled Breath Test for the Diagnosis of Oesophagogastric Cancer. JAMA Oncol. 2018 Jul 1;4(7):970-976. doi: 10.1001/jamaoncol.2018.0991. PMID 29799976